CLINICAL TRIAL: NCT03841201
Title: IMMUNIB - An Open-label, Single-arm Phase II Study of Immunotherapy With Nivolumab in Combination With Lenvatinib for Advanced Stage Hepatocellular
Brief Title: Immunotherapy With Nivolumab in Combination With Lenvatinib for Advanced Stage Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Collaborators: Bristol-Myers Squibb (Industry); Eisai GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMMUNIB
Record Dates: First submitted 2019-02-12; First posted 2019-02-15 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib; Pharmaceutical Preparations; Nivolumab

STUDY DESIGN:
Intervention Model Description: Open-label, single-arm, multicenter phase II trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): * Lenvatinib peroral qd (8 mg for patients with body weight <60kg and 12 mg for patients with body weight ≥ 60kg)
  * Nivolumab i.v. q2w (240mg fixed dose IV) max. 36 cycles
  Interventions: Drug: Lenvatinib; Drug: Nivolumab

INTERVENTIONS:
Drug: Lenvatinib — oral
  Other Names: Study treatment
Drug: Nivolumab — iv infusion
  Other Names: Study treatment

SUMMARY:
This is an exploratory, open-label, single arm, multicenter phase II trial for the evaluation of efficacy and feasibility (as determined by safety and tolerability) of immunotherapy with nivolumab in combination with lenvatinib for patients with multinodular, advanced stage hepatocellular carcinoma in first line therapy

ELIGIBILITY:
Inclusion Criteria:

1. Fully-informed written consent.
2. Males and females ≥ 18 years of age

   *There are no data that indicate special gender distribution. Therefore patients will be enrolled in the study gender-independently.
3. Unresectable, multinodular tumour, not eligible for resection or local ablation
4. Histologically confirmed diagnosis of hepatocellular carcinoma
5. Has a Child-Pugh Classification score ≤ 6 for assessed liver function within 7 days before allocation (Appendix 4: Child-Pugh Score)
6. At least one measurable site of disease as defined by RECIST 1.1 criteria with spiral CT scan or MRI.
7. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.
8. Life expectancy of at least 12 weeks.
9. Adequate bone marrow, hepatic and renal function including the following:

   * Haemoglobin ≥ 10.0 g/dL, absolute neutrophil count ≥ 1,500 /µL, platelets ≥70,000 /µL;
   * Total bilirubin ≤ 3.0 mg/dL upper normal limit;
   * AST (SGOT), ALT (SGPT) ≤ 5 x upper normal limit;
   * International normalized ratio (INR) ≤1.25;
   * Albumin ≥ 30 g/dL;
   * Creatinine ≤ 1.5 x upper normal limit OR measured or calculated creatinine clearance (according to Cockcroft-Gault) ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN (GFR can also be used in place of creatinine or CrCl)
10. Female patients with reproductive potential must have a negative urine or serum pregnancy test within 7 days prior to start of trial. Women must not be breastfeeding.
11. If patient has concurrent Hepatitis B virus (HBV) or Hepatitis C virus (HCV) infection, meets the following criteria:

    * Patients with HBV or HCV infection should be monitored for viral levels during study participation.
    * Patients with detectable hepatitis B surface antigen (HBsAg) or detectable HBV DNA should have HBV DNA < 100 IU/ml and should be managed per local treatment guidelines.

    Controlled (treated) hepatitis B subjects will be allowed if they started treatment at the time point of enrollment into the study by the latest and treatment is continued during study participation and for ≥ 6 months after end of study treatment.

    - HCV patients with with advanced HCC are mostly not treated for their HCV infection. However, patients treated for HCV are considered suitable for inclusion if antiviral therapy has been completed ≥ 30 days prior to first administration of study drug.
12. The patient is willing and able to comply with the protocol for the duration of the study, including hospital visits for treatment and scheduled follow-up visits and examinations.
13. WOCBP must agree to follow instructions for method(s) of contraception for a period of 30 days (duration of ovulatory cycle) plus the time required for the investigational drug to undergo 5 half-lives. The terminal half-lives of nivolumab is approximately 25 days. WOCBP should use an adequate method to avoid pregnancy for approximately 5 months (30 days plus the time required for nivolumab to undergo 5 half-lives) after the last dose of investigational drug.
14. Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for a period of 90 days (duration of sperm turnover) plus the time required for the investigational drug to undergo 5 half-lives. The terminal half-lives of nivolumab is approximately 25 days. Males who are sexually active with WOCBP must continue contraception for approximately 7 months (90 days plus the time required for nivolumab to undergo 5 half-lives) after the last dose of investigational drug. In addition, male subjects must be willing to refrain from sperm donation during this time.

Exclusion Criteria:

1. Previous systemic therapy in the first-line setting.
2. Patients on a liver transplantation list or with advanced liver disease as defined below:

   * Encephalopathy
   * Untreatable Ascites.
3. Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC.
4. Prior organ allograft or allogeneic bone marrow transplantation.
5. Local therapies ongoing or completed <4 weeks prior to the baseline scan.
6. Thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within the 6 months prior to the first dose of study drug with the exception of thrombosis of a segmental portal vein.
7. Prior, systemic anti-cancer chemotherapy, radiotherapy administered <4 weeks prior to study entry, endocrine- or immunotherapy or use of other investigational agents.
8. History of (non-infectious) pneumonitis that required steroids or current pneumonitis.
9. Major surgery within 4 weeks of starting the study. Patients must have recovered from effects of major surgery.
10. Malignancies other than disease under study within 5 years prior to inclusion, with the exception of those with a negligible risk of metastasis or death (e.g., expected 5-year OS > 90%) treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, ductal carcinoma in situ treated surgically with curative intent)
11. Uncontrolled hypertension.
12. Clinically significant cardiovascular disease.
13. Any serious or uncontrolled medical disorder or active infection that, in the opinion of the investigator, may increase the risk associated with study participation, study drug administration, or would impair the ability of the subject to receive study drug.
14. Proteinuria (≥2g/24h)
15. Psychiatric disorders or altered mental status precluding understanding of the informed consent process and/or compliance with the study protocol.
16. Subjects with a history of or current CNS metastases. A scan to confirm the absence of brain metastases is not required. Patients with unknown CNS metastatic status and any clinical signs indicative of CNS metastases are eligible if CNS metastases are excluded using CT and/or MRI scans.
17. Pregnant or breast-feeding women.
18. Immunocompromised patients, e.g. patients who are known to be serologically positive for human immunodeficiency virus (HIV).
19. Subjects with active, known, or suspected autoimmune disease. Subjects with Type I diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement, or skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment are permitted to enroll. For any cases of uncertainty, it is recommended that the medical monitor be consulted prior to signing informed consent.
20. Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids, and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
21. Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
22. All toxicities attributed to prior anti-cancer therapy other than hearing loss, alopecia and fatigue must have resolved to Grade 1 (NCI CTCAE version 4.03) or baseline before administration of study drug.
23. > Grade 1 peripheral neuropathy according to CTCAE version 4.03
24. Patients who have received a live vaccine within 30 days prior to enrolment.
25. History of allergy or hypersensitivity to study drugs or any constituent of the products
26. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.
27. Patient who has been incarcerated or involuntarily institutionalized by court order or by the authorities § 40 Abs. 1 S. 3 Nr. 4 AMG.
28. Patients who are unable to consent because they do not understand the nature, significance and implications of the clinical trial and therefore cannot form a rational intention in the light of the facts [§ 40 Abs. 1 S. 3 Nr. 3a AMG].

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) according to RECIST 1.1 | 6 months
  Number and percentage of participants with a best overall response (BOR) of complete response (CR) or partial response (PR) according to RECIST 1.1
Safety and tolerability (AEs, SAEs according to NCI-CTCAE V 4.03) | 6 months
  Type, incidence and severity of AEs, SAEs according to NCI-CTCAE V 4.03

SECONDARY OUTCOMES:
Objective response rate (ORR) according to iRECIST | 6 months
  Number and percentage of participants with a best overall response (BOR) of complete response (CR) or partial response (PR) according to iRECIST
Time-to-progression (TTP) | 6 months
  Time from the date of treatment allocation to the date of first observed disease progression (investigator assessment according to RECIST 1.1).
Progression free survival (PFS) | 6 months
  Time from the date of treatment allocation to the date of first observed disease progression (investigator assessment according to RECIST 1.1) or death from any cause.
Overall survival (OS) | 6 months
  Time from the date of treatment allocation to the date of death (due to any cause).
Translational research | 6 months
  Correlation of biomarkers potentially associated with clinical efficacy (OS, PFS and ORR) from lenvatinib plus nivolumab by molecular quantitation of mRNA expression of parameters like e.g. PD-1, PD-L1 and PD-L2, immune cell infiltrates (IGHM, CD3, CD8, FOXP3, CD68, CD205), chemokines (CXCL9, CXCL10, CXCL13) and invasion markers (MMP7, MMP9).

CONTACTS AND LOCATIONS:
Overall Officials: Salah-Eddin Al-Batran, MD, Study Director — Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest
Locations (1):
- Hannover Medical School, Hanover, Germany

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared